CLINICAL TRIAL: NCT01633580
Title: Follicular Phase Endocrine Characteristics During Ovarian Stimulation and GnRH Antagonist Co-treatment for IVF; Randomized Trial Comparing Corifollitropin Alfa (Elonva) Initiated on Cycle Day 2 or 4.
Brief Title: D2 Versus D4 Corifollitropin Alfa in GnRH Antagonists
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Blockeel Christophe, MD, PhD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/019
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
Keywords: ICSI; GnRH antagonist; corifollitropin alfa
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 2 group (Placebo Comparator): Patients undergo a standard treatment with a classical start of corifollitropin alfa in a GnRH antagonist protocol.
  Interventions: Drug: corifollitropin alfa
- Day 4 group (Active Comparator): Patients undergo an ovarian stimulation, but start on day 4 with corifollitropin alfa
  Interventions: Drug: corifollitropin alfa

INTERVENTIONS:
Drug: corifollitropin alfa — long acting FSH

SUMMARY:
The purpose of the present study is to analyse if corifollitropin alfa, an agent for prolonged ovarian stimulation, administered from day 4 can be clinically used instead of day 2 onwards for a controlled ovarian hyperstimulation (COH) in an antagonist protocol.

DETAILED DESCRIPTION:
Corifollitropin alfa is a new recombinant gonadotrophin with sustained follicle-stimulating activity. It offers novel and effective treatment option for potential normal responder patients undergoing ovarian stimulation with GnRH antagonist co-treatment for IVF or in vitro fertilisation resulting in a high ongoing pregnancy rate, equal to that achieved with daily rFSH. Normally, this medication is started on day 2 of the cycle. In the present randomised trial, we want to evaluate whether this agent can be clinically used when started on day 4 of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* < 36 years old on day of randomisation
* FSH < 12 (in the early follicular phase)
* Normal ultrasound scan, i.e. presence of both ovaries, without evidence of abnormality within 6 months prior to randomisation.
* Regular menstrual cycles of 21-35 days, presumed to be ovulatory.
* BMI ≤ 29
* Weight > 60 kg
* < 3 previous trials
* ICSI
* Randomisation at out-patient clinic

Exclusion Criteria:

* ≥ 36 years old on day of randomisation
* Endometriosis ≥ grade 3
* PCOS
* Poor responders (development of < 4 follicles in a previous IVF/ICSI cycle)
* Endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney)

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Consumption of rFSH at the end of the follicular phase | up to 9 months
  The purpose is to assess the additional need for recFSH in each treatment group

SECONDARY OUTCOMES:
Pregnancy rate | Up to 9 months
  The purpose is to study the pregnancy rate in each treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

REFERENCES:
- [Derived] Blockeel C, Polyzos NP, Derksen L, De Brucker M, Vloeberghs V, van de Vijver A, De Vos M, Tournaye H. Administration of corifollitropin alfa on Day 2 versus Day 4 of the cycle in a GnRH antagonist protocol: a randomized controlled pilot study. Hum Reprod. 2014 Jul;29(7):1500-7. doi: 10.1093/humrep/deu105. Epub 2014 May 9. PMID 24813196